CLINICAL TRIAL: NCT03395548
Title: Stability of the Intestinal Microbiome in Patients Suffering From Inflammatory Bowel Disease (IBD) and Irritable Bowel Syndrome (IBS) Under the Influence of an Osmotic Laxans
Brief Title: Stability of the Microbiome in IBD and IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 29-255 ex 16/17
Record Dates: First submitted 2017-11-14; First posted 2018-01-10 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Microbiota
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inflammatory bowel disease (Active Comparator): The aim is to recruit 20 persons suffering from Crohn's disease or ulcerative colitis with stable medication and stable control of the disease.
  As in each group the intervention will be the colon lavage with macrogol in combination with the colonoscopy.
  Interventions: Drug: Macrogol
- Irritable bowel syndrome (Active Comparator): The aim is to recruit 20 persons suffering from irritable bowel syndrome (IBS) fulfilling rome criteria.
  As in each group the intervention will be the colon lavage with macrogol in combination with the colonoscopy.
  Interventions: Drug: Macrogol
- Healthy (Active Comparator): The aim is to recruit 20 persons without known illnesses with a comparable age to the other two groups.
  As in each group the intervention will be the colon lavage with macrogol in combination with the colonoscopy.
  Interventions: Drug: Macrogol

INTERVENTIONS:
Drug: Macrogol — Used drug: Macrogol (osmotic laxative)

SUMMARY:
In this study the investigators aim to investigate the changes of the intestinal microbiome in three different cohorts (IBD, IBS, healthy) after applying the uniform disruptive factor of osmotic diarrhea induced by macrogol. The investigators hypothesis is that ill people will show more severe changes of the microbiome than healthy people and that these changes persist longer.

DETAILED DESCRIPTION:
I

ELIGIBILITY:
Inclusion Criteria:

* patients with inflammatory bowel disease and irritable bowel syndrome and stable therapy since three months
* patients with the indication for colonoscopy

Exclusion Criteria:

* age under 18
* pregnancy
* new therapy planned
* change of therapy within the last three months
* acute exacerbation of the inflammatory bowel disease
* colon pathologies of other origin: colocarcinoma, Illnesses with diarrhea (f.e.microscopic colitis), short bowel syndrome, malabsorption, colectomy
* intake of antibiotics in the last three months
* intake of probiotics in the last month
* intake of antibiotics or probiotics during the study
* new proton pump inhibitor therapy
* significant change of nutrition in the last three months
* holidays outside europe in the last month
* gastroenteritis in the last three months
* intake of laxatives
* nonsteroidal antiinflammatory drugs should be avoided and documented

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Changes of the microbiome | 4 months
  The investigators aim to asses the changes of the gut microbiome between the three Groups and before and after lavage (Alpha Diversity, Beta Diversity, Group Significance)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Blesl, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Universitätsklinikum Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided